CLINICAL TRIAL: NCT06115707
Title: Head Positioning After Endovascular Therapy for Acute Ischemic Stroke: A Randomized Controlled Trial
Brief Title: Head Position After Endovascular Therapy
Acronym: HeadSOAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou Yuan (Other)
Responsible Party: Sponsor-Investigator, Zhengzhou Yuan, MD, The Affiliated Hospital Of Southwest Medical University
Organization: The Affiliated Hospital Of Southwest Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SWMU202305
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Stroke, Acute; Endovascular Therapy
MeSH Terms: conditions — Stroke | interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The lying flat group (Active Comparator): Patients in lying flat intervention to be nursed lying flat (0°-10°) after endovascular therapy is made and to remain in this position for 72 hours.
  Interventions: Other: The lying flat (0°-10°) head position for 72 hours
- The head elevation group (Experimental): Patients in the sitting up intervention should be nursed with their head elevated (30°-40°) by raising the head of the bed (or using extra pillows or wedges) after undergoing endovascular therapy, and to remain in this position for 72 hours.
  Interventions: Other: The The head elevation (30°-40°) position for 72 hours

INTERVENTIONS:
Other: The lying flat (0°-10°) head position for 72 hours — The lying flat (0°-10°) head position for 72 hours after endovascular therapy.
  Arms: The lying flat group
Other: The The head elevation (30°-40°) position for 72 hours — The head elevoatin (30°-40°) position for 72 hours after endovascular therapy.
  Arms: The head elevation group

SUMMARY:
The aim of this trial is to investigate whether head elevation position after endovascular treatment can improve the 90-day functional outcome of acute large vessel occlusion in the anterior circulation.

DETAILED DESCRIPTION:
The optimal head position for patients with acute ischemic stroke (AIS) remains uncertain. The HeadPoS study revealed that there is no significant difference in disability outcomes between patients who are placed in a lying-flat position for 24 hours and those who are placed in a sitting-up position with the head elevated to at least 30 degrees for 24 hours. However, this study included both patients with ischemic and hemorrhagic strokes, and most of the patients had mild strokes (median National Institutes of Health Stroke Scale score of 4). It is unclear how to arrange the patient's head position after endovascular treatment.

The hypothesis of this trial: Compared with the lying flat head positioni, the head elevation position after endovascular treatment can significantly improve the 90-day functional outcome of acute large vessel occlusion in the anterior circulation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs consistent with acute ischemic stroke;
2. Age ≥ 18 years old;
3. Proved anterior circulation large vessel occlusion on digital subtraction angiography (ICA, M1, M2) with/without cervical lesion (tandem);
4. NIHSS score ≥ 8 points before endovascular treatment;
5. ASPECTS score ≤ 7 points before endovascular treatment;
6. Successful vessel recanalization after endovascular treatment (defined as an eTICI score of 2b, 2c, or 3) ；
7. The time from onset to randomization ≤ 24 hours (the onset time is defined as the last normal time);
8. Written informed consent is obtained from patients and/or their legal representatives.

Exclusion Criteria:

1. Pre-stroke mRS score>1 point;
2. Patients with acute occlusions in multiple vascular territories (e.g. bilateral anterior circulation, or anterior/posterior circulation);
3. Currently in pregnant or lactating or serum beta HCG test is positive on admission;
4. Contraindications to a flat head position;
5. Any terminal illness with life expectancy less than 6 months;
6. Participating in other clinical trials;
7. Patients with a preexisting neurological or psychiatric disease that would confound the neurological functional evaluations;
8. Unlikely to be available for 90-day follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1368 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2025-04-26 (Actual)

PRIMARY OUTCOMES:
Modified Rankin scale score (mRS) | 90 days
  disability level. The presence of impairments determines the transitions from mRS score 0 to mRS score 1 (symptoms) and mRS score 5 to mRS score 6 (death).

SECONDARY OUTCOMES:
Proportion of patients non-disabled (mRS score 0 to 1) or return to pre-morbid mRS score at 90 days (for patients with mRS > 1) | 90 days
  excellent outcome
Proportion of patients functionally independent (mRS score 0 to 2) at 90 days | Within 90 days90 days
  functional independence
Proportion of patients ambulatory or bodily needs-capable or better (mRS score 0 to 3) | 90 days
  ambulatory or bodily needs-capable or better
Health-related quality of life, assessed with the EuroQol-visual analogue scales (EQ-VAS) | 90 days
  Health-related quality of life
Mortality within 90 days | 90 days
  evaluate death rate of the two treatment groups
severe adverse events | within 90 days
  evaluate complications and any adverse events
Symptomatic intracerebral hemorrhage incidence (Heidelberg Criteria) | within 72 hours after randomized
  evaluate intracranial hemorrhage
Any type of intracerebral hemorrhage (Heidelberg Criteria) | within 72 hours after randomized
  evaluate intracranial hemorrhage
Brain edema | within 72 hours after randomized
  evaluate brain edema
Malignant Brain Edema | within 72 hours after randomized
  evaluate brain edema
Incidence of pulmonary infections | within 72 hours after randomized
  evaluate pulmonary infections
Improvement in National Institute of Health stroke scale (NIHSS) score between baseline and 5~7d | at 5~7 days after randomization
  neurological changes.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengzhou Yuan, Study Chair — Affiliated Hospital of Southwest Medical University; Yong Jiang, Study Chair — Affiliated Hospital of Southwest Medical University
Locations (67):
- China (67):
  - Chongqing Banan District People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Bishan District People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Ninth People's Hospital, Chongqing, Chongqing Municipality
  - Yongchuan Hospital Affiliated to Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Longyan First Hospital, Longyan, Fujian
  - Dingxi People's Hospital, Dingxi, Gansu
  - Jiuquan People's Hospital, Jiuquan, Gansu
  - Gansu Provincial Hospital of Traditional Chinese Medicine, Lanzhou, Gansu
  - Lanzhou University First Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Tianshui First People's Hospital, Tianshui, Gansu
  - Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong
  - Guangdong Provincial People's Hospital Heyuan Hospital, Heyuan, Guangdong
  - Baise People's Hospital, Baise City, Guangxi
  - Nanning Third People's Hospital, Nanning, Guangxi
  - Qiannan Prefecture People's Hospital, Duyun, Guizhou
  - Xingyi People's Hospital, Xingyi, Guizhou
  - The First Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - Jiamusi Central Hospital, Jiamusi, Heilongjiang
  - Yichun First Hospital, Yichun, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Xihua County People's Hospital, Zhoukou, Henan
  - Shiyan taihe hospital, Shiyan, Hubei
  - Ningxiang First People's Hospital, Changsha, Hunan
  - The First People's Hospital of Chenzhou City, Chenzhou, Hunan
  - Ganzhou Municipal Hospital, Ganzhou, Jiangxi
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Xingguo County People's Hospital, Ganzhou, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Dalian 967 Hospital, Dalian, Liaoning
  - Ningxia Hui Autonomous Region People's Hospital, Yinchuan, Ningxia
  - The Fifth People's Hospital of Qinghai Province, Xining, Qinghai
  - Baoji High tech Hospital, Baoji, Shaanxi
  - Northwest University Affiliated Hospital, Xi'an, Shaanxi
  - Xidian Group Hospital, Xi'an, Shaanxi
  - Xianyang First People's Hospital, Xianyang, Shaanxi
  - Yulin First Hospital, Yulin, Shaanxi
  - Rizhao Traditional Chinese Medicine Hospital, Rizhao, Shandong
  - Shanxi Provincial Hospital, Taiyuan, Shanxi
  - Chengdu Sixth People's Hospital, Chengdu, Sichuan
  - Chongzhou People's Hospital, Chengdu, Sichuan
  - Deyang People's Hospital, Deyang, Sichuan
  - Guangyuan First People's Hospital, Guangyuan, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Gulin County People's Hospital, Luzhou, Sichuan
  - Beichuan County People's Hospital, Mianyang, Sichuan
  - Mianyang 404 Hospital, Mianyang, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Neijiang Second People's Hospital, Neijiang, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Suining First People's Hospital, Suining, Sichuan
  - Liangshan First People's Hospital, Xichang, Sichuan
  - Xichang People's Hospital, Xichang, Sichuan
  - Ya'an People's Hospital, Ya'an, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Fushun County People's Hospital, Zigong, Sichuan
  - Zigong First People's Hospital, Zigong, Sichuan
  - Zigong Fourth People's Hospital, Zigong, Sichuan
  - Zigong Third People's Hospital, Zigong, Sichuan
  - The Seventh Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Qujing First People's Hospital, Qujing, Yunnan
  - Wenzhou Medical University First Affiliated Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No